CLINICAL TRIAL: NCT04288362
Title: The Patient Activation Through Community Empowerment/Engagement for Diabetes Management (PACE-D) Protocol: A Non-randomised Controlled Trial of Personalised Care and Support Planning for Persons Living With Diabetes
Brief Title: Patient Activation Through Community Empowerment/Engagement for Diabetes Management (PACE-D)
Acronym: PACE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Tan Wee Hian, PACE-D Programme Director, Consultant Family Physician, National University Health System, Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-SN-03
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus; Chronic Disease; Patient Care Planning; Patient Participation; Self Care; Empowerment
Keywords: Diabetes; Long term conditions; Chronic disease management; Patient engagement; Patient empowerment; Self-management; Care Planning
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease; Patient Participation; Empowerment | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Non-randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Intervention Group
- Control Group (Active Comparator)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group — Participants in this arm will undergo the new care model for management of diabetes mellitus polyclinics.
  Arms: Intervention Group
Other: Control Group — Participants in this arm will continue to undergo the existing care model for management of diabetes mellitus in the polyclinics.
  Arms: Control Group

SUMMARY:
The study is a non-randomised controlled trial involving an intervention group and a control group. It aims to evaluate the effects of a patient engagement and empowerment model of collaborative care support planning on clinical outcomes of patients with diabetes mellitus as compared to usual care in the primary care setting. It also aims will be to examine the impact of the intervention on patient activation, patient and healthcare provider experience, and healthcare utilisation.

DETAILED DESCRIPTION:
The investigators will conduct a prospective study on existing patients with diabetes who are on follow-up with their teamlets at Pioneer (PIO), Jurong (JUR), Bukit Batok (BBK) and Choa Chu Kang (CCK) polyclinics for management of diabetes. Recruitment will occur for 18 months from the time of study implementation. One teamlet in JUR and one teamlet in PIO (total of two teamlets) will fall under intervention arm where the new care model based on the Year-of-Care (YOC) model will be delivered, whereas one teamlet in BBK and one teamlet in CCK (total of another two teamlets) will fall under the control arm where the current teamlet model will be continued.

In the intervention group, patients recruited will undergo the new care model which entails receiving the Care Planning Results Letter before the consultation at their annual review, involving them in the Care and Support Planning (CSP) consultation at the annual review, and referring them to suitable community resources to support self-management. The Care Planning Results Letter prompts patients to think the issues they would like to raise to their Doctor or Care Manager (who is a nurse trained in chronic disease management), checks on their mood, provides information on their most recent few laboratory test results, clinical parameters, smoking status, and attendances for foot and eye screenings. The letter also covers goal setting and action planning discussions. The patient is expected to bring it for the upcoming CSP consultation at the annual review. The CSP is a conversation which is conducted by the Doctor or Care Manager trained in the new care model. It focuses on a collaborative approach between the health care providers and the patient for joint goal setting and shared decision making to support self-management of their chronic condition(s).

In the control arm, the participants will receive the usual care with the teamlet model. There will not be any Care Planning Results Letter prepared for the patient. At the upcoming annual visit, the patient will continue to have the usual annual review for the laboratory test results and consultation. A flyer that lists the community programmes that support the patient for self-management will also be issued to the patient. If the patient is interested in any of these programmes, they may sign up with the respective community providers directly.

After the first CSP, selected patient participants may be invited for a one-to-one in-depth interviews (IDIs) to explore their perceptions about diabetes, diabetes management and the intervention programme in greater detail. The interviews will be conducted by researchers trained qualitative research methodology. They will be semi-structured with a topic guide to support exploration of the themes of interest, and will be informed by prior qualitative research with this and other similar interventions, as well as the results from the patient surveys. Health care providers who are involved in the delivery of CSPs in the intervention arm will also be invited for a one-to-one in-depth interviews (IDIs), to develop an understanding of how they find the training and new way of working with patients (particularly the care and support planning conversation).

ELIGIBILITY:
Inclusion Criteria:

* On follow up with an existing teamlet pre-assigned to participate in the study
* Adults with diabetes mellitus
* Age 21 years and above
* Ability to provide informed consent
* Ability to communicate in the language(s) which the physician is confident to carry out the care and support planning consult in English, Malay or Chinese
* Ability to read and comprehend the Diabetes Results Letter on their own OR has family members who are able to assist to that

Exclusion Criteria:

* Doctors, Care Managers and Care Coordinators involved in the care and support planning process
* Age 21 years and above
* Ability to provide informed consent

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1620 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels | From baseline to study endpoint, one year in general
  Change in HbA1c levels in patients receiving the CSP intervention compared with patients receiving standard care.

SECONDARY OUTCOMES:
Change in mean Patient Activation Measures-13 (PAM-13) scores | From baseline to study endpoint, one year in general
  Change in mean Patient Activation Measures-13 (PAM-13) scores in patients receiving the CSP intervention compared with patients receiving standard care. PAM-13 is a validated tool with 13-item response rated on a 4-point Likert-type scale that will be converted to a linear score of 0 (lowest patient activation) to 100 (highest patient activation). Higher patient activation score from PAM-13 is associated better healthcare outcomes such as medication adherence.
Change in proportion of patients in the various ranges of patient activation levels | From baseline to study endpoint, one year in general
  Change in proportion of patients in the various ranges of patient activation levels for patients receiving the CSP intervention compared with patients receiving standard care.
Change in healthcare utilisation in terms of number of polyclinic visits | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of number of polyclinic visits for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare utilisation in terms of proportion (%) of patients with emergency department visits | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of proportion (%) of patients with emergency department visits for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare utilisation in terms of number of emergency department visits | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of number of emergency department visits for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare utilisation in terms of proportion (%) of patients with hospital inpatient admissions | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of proportion (%) of patients with hospital inpatient admissions for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare utilisation in terms of number of hospital inpatient admissions | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of number of hospital inpatient admissions for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare utilisation in terms of proportion (%) of patients with specialist outpatient clinic visits | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of proportion (%) of patients with specialist outpatient clinic visits for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare utilisation in terms of number of specialist outpatient clinic visits | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare utilisation in terms of number of specialist outpatient clinic visits for patients receiving CSP intervention compared with patients receiving standard care, assessed through retrospective analysis of electronic medical records.
Change in healthcare cost in terms of total healthcare cost of polyclinic, emergency department, hospital admissions and specialist outpatient clinic visits | Two years in general from one year preceding recruitment to the period between first and second annual reviews
  Change in healthcare cost in terms of total healthcare cost of polyclinic, emergency department, hospital admissions and specialist outpatient clinic visits in patients receiving the CSP intervention compared with patients receiving standard care.

OTHER OUTCOMES:
Change in proportion of patients meeting their target blood pressure levels | From baseline to study endpoint, one year in general
  Change in proportion of patients meeting their target blood pressure levels for patients receiving the CSP intervention compared with patients receiving standard care.
Change in proportion of patients meeting their target LDL-cholesteterol levels | From baseline to study endpoint, one year in general
  Change in proportion of patients meeting their target LDL-cholesteterol levels for patients receiving the CSP intervention compared with patients receiving standard care.
Change in body weight | From baseline to study endpoint, one year in general
  Change in body weight (kg) in patients receiving the CSP intervention compared with patients receiving standard care.
Change in exercise duration | From baseline to study endpoint, one year in general
  Change in exercise duration (minutes per week) in patients receiving the CSP intervention compared with patients receiving standard care.
Change in smoking rates | From baseline to study endpoint, one year in general
  Change in smoking rates (cigarettes per day) in patients receiving the CSP intervention compared with patients receiving standard care.
Change in the proportion (%) of patients who indicate community resource utilisation | From baseline to study endpoint, one year in general
  Change in the proportion (%) of patients who indicate community resource utilisation in the past 1 year between patients CSP intervention compared with patients receiving standard care. Community resource utilisation history is assessed through dichotomous questionnaire with yes/no response.
Change in Diabetes Foot Screening rates | From baseline to study endpoint, one year in general
  Change in Diabetes Foot Screening Rates in patients receiving the CSP intervention compared with patients receiving standard care.
Change in Diabetes Retinal Photography rates | From baseline to study endpoint, one year in general
  Change in Diabetes Retinal Photography rates in patients receiving the CSP intervention compared with patients receiving standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Young, Study Chair — National University Health System, Singapore; Victor Weng Keong Loh, Study Director — National University Health System, Singapore; Tong Wei Yew, Study Director — National University Hospital, Singapore; Kavita Venkataraman, Study Director — National University of Singapore; Brent Gibbons, Study Director — National University of Singapore; Vikki Entwistle, Study Director — National University of Singapore; Soon Guan Tan, Study Director — National University of Singapore; Meena Sundram, Study Director — National University Health System, Singapore; Keith Tsou, Study Director — National University Health System, Singapore; Yii Jen Lew, Study Director — National University Health System, Singapore; Wee Hian Tan, Principal Investigator — National University Health System, Singapore
Locations (1):
- National University Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coulter A, Entwistle VA, Eccles A, Ryan S, Shepperd S, Perera R. Personalised care planning for adults with chronic or long-term health conditions. Cochrane Database Syst Rev. 2015 Mar 3;2015(3):CD010523. doi: 10.1002/14651858.CD010523.pub2. PMID 25733495
- [Background] Wagner EH, Austin BT, Von Korff M. Organizing care for patients with chronic illness. Milbank Q. 1996;74(4):511-44. PMID 8941260
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Derived] Tan WH, Loh VWK, Venkataraman K, Choong ST, Lew YJ, Sundram M, Tsou K, Tan SG, Gibbons B, Entwistle V, Young D, Tai ES, Yew TW. The Patient Activation through Community Empowerment/Engagement for Diabetes Management (PACE-D) protocol: a non-randomised controlled trial of personalised care and support planning for persons living with diabetes. BMC Fam Pract. 2020 Jun 19;21(1):114. doi: 10.1186/s12875-020-01173-2. PMID 32560689